CLINICAL TRIAL: NCT07089004
Title: Co-relation of Hypomagnesemia With Clinical Outcomes in Critically Ill Patients Admitted to a Tertiary Care ICU in Bangladesh
Brief Title: Hypomagnesemia and Its Clinical Outcome
Acronym: Hypogamnesamia
Status: Completed | Type: Observational
Sponsor: Bangladesh Bioscience Research Group (Network)
Collaborators: Chattogram International Dental College (Other); Chittagong Medical College and Hospital (Other); Bangladesh Medical University (Other)
Responsible Party: Principal Investigator, Pair Ahmed Jiko, Lab-Incharge (Biochemist), Bangladesh Medical Research Council (BMRC)
Other Study IDs: BBMH/2023/RP-2342; BBMH/June/2023/011 (Registry Identifier: Institute of Applied Health Sciences-USTC (ex-Bangabandu Memorial Hospital))
Record Dates: First submitted 2025-06-29; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Hypomagnesemia; Critical Illness; Intensive Care Unit (ICU) Patients; Scoring Systems
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood: Serum/Plasma Samples were collected from critically ill patients admitted to the Intensive Care Unit (ICU). The retained biospecimen will include serum samples, which will be used to measure serum magnesium levels and other relevant biochemical parameters as part of routine clinical assessment and research analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: No intervention (observational study) — Observational - Biochemical, Hematological and Clinical Scoring Assessments

SUMMARY:
Magnesium is an essential electrolyte involved in numerous physiological processes, including maintaining cellular integrity, regulating muscle tone, supporting cardiovascular function, and modulating immune responses. Despite its critical role, magnesium is often overlooked in clinical practice, earning it the title of the "forgotten electrolyte." Hypomagnesemia, defined as serum magnesium levels below 1.5 mEq/L, has been associated with adverse clinical outcomes such as increased mortality, prolonged ICU stays, and higher requirements for mechanical ventilation. Critically ill patients are particularly vulnerable to hypomagnesemia due to various underlying conditions, gastrointestinal losses, and renal complications. However, limited data are available from Bangladesh on the burden and clinical impact of hypomagnesemia in ICU settings. This study aims to assess the correlation between hypomagnesemia and clinical outcomes, including length of ICU stay, need for mechanical ventilation, and mortality among critically ill patients in a tertiary care ICU in Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above.
* Patients admitted to the Intensive Care Unit (ICU).
* Patients who have serum magnesium levels measured within 24 hours of ICU admission.

Exclusion Criteria:

* Patients with known end-stage renal disease on dialysis.
* Patients with a history of magnesium supplementation prior to ICU admission.
* Pregnant women.
* Patients with incomplete medical records or unavailable laboratory data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will consist of critically ill adult patients admitted to the Intensive Care Unit (ICU) of a tertiary care hospital in Bangladesh. The study will include both male and female patients aged 18 years and above, irrespective of their underlying diagnosis, provided they meet the inclusion criteria. Patients will be assessed for serum magnesium levels (Hypo; Normo and Hyper) within 24 hours of ICU admission, along with relevant biochemical, hematological and clinical parameters. The study will exclude individuals with known end-stage renal disease on dialysis, those receiving magnesium supplementation prior to ICU admission, pregnant women and patients with incomplete medical records.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Association of Hypomagnesemia with ICU Mortality | From the date of ICU admission until the date of ICU discharge or death, assessed up to 60 days.
  To assess the relationship between low serum magnesium levels and all-cause mortality among critically ill ICU patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Science and Technology Chittagong (USTC), Chittagong, Khulshi, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared with other researchers to ensure the protection of patient confidentiality and comply with institutional and ethical guidelines. Only aggregated, de-identified data may be shared upon reasonable request and with appropriate ethical approvals.